CLINICAL TRIAL: NCT05559658
Title: A Cross-sectional Descriptive Study Using Mixed Method (Qualitative and Quantitative) Data Collection
Brief Title: Comprehensive Assessment in a Longitudinal Study on Young Men Who Have Sex With Men Attracting to chemseX
Acronym: CLYMAX
Status: Recruiting | Type: Observational
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Other Study IDs: IHRI021
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: ChemSex Users for YMSM; ChemSex Users
Keywords: ChemSex users

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: A: Current chemsex users Men who have sex with men, Aged 16-35 years, Able to communicate in Thai fluently, Current chemsex users.
  B: Former chemsex users (discontinued ≥90 days) Men who have sex with men, Aged 16-35 years, Able to communicate in Thai fluently, Former chemsex users (discontinued ≥90 days).

SUMMARY:
The study is a two-phase observational study that assess multiple aspects of study and young men who have sex with men (YMSM).

Phase I of the study will be a cross-sectional descriptive study using a mixed methods data collection (focusing on qualitative data collection) to acquire information necessary for developing a more extensive study on the same matter.

Phase II of the study will be a prospective cohort study using a quantitative data collection.

Findings from phase I will guide the development of phase II which consist of a larger number of YMSM, important baseline and follow-up questionnaires and comorbidities assessments, sexually transmitted infections testing, and integration to care.

This protocol exclusively addresses the phase I of the study.

Once the phase I findings are finalized, the principal investigator will submit the phase II to the IRB of the Faculty of Medicine, Chulalongkorn University.

ELIGIBILITY:
Inclusion Criteria:

Group 1A: Current chemsex users

1. Men who have sex with men
2. Aged 16-35 years
3. Able to communicate in Thai fluently
4. Current chemsex users
5. Provide informed consent

Inclusion Criteria:

Group 1B: Former chemsex users (discontinued ≥90 days)

1. Men who have sex with men
2. Aged 16-35 years
3. Able to communicate in Thai fluently
4. Former chemsex users (discontinued ≥90 days)
5. Provide informed consent

Exclusion Criteria:

No exclusion criteria for all groups of participants

Ages: 16 Years to 35 Years | Sex: Male
Age Groups: Child, Adult
Study Population: Current chemsex users
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The study will be divided into two phases. The information on the procedures of the phase I single study visit is presented below. | 12 months
  Qualitative data collection The qualitative study component will use semi-structured individual in-depth interviews (IDIs) in Thai conducted in-person at the team community health clinic facilities. All participants will be included in the qualitative data collection - 40 YMSM, all 10 family members or peers of chemsex users, and all 10 clinic staff.
  Quantitative data collection Demographic information of all participants, the proportion of all eligible participants who agree to participate in the study, and the relationship status between Group 2 and Group 1 participants will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of HIV Research and Innovation, Pathum Wan, Bangkok, Thailand